CLINICAL TRIAL: NCT04393974
Title: OnCovid: Natural History and Outcomes of Cancer Patients During the COVID19 Epidemic
Brief Title: COVID-19 and Cancer Patients
Acronym: OnCovid
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 282140
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Sars-CoV2
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients with COVID-19: All cancer patients can be recruited onto this research following a positive test for Sars-Cov2. The research will follow what treatments they are given for the infection, but also look at their past medical history including prior and any current anti-cancer therapy.

SUMMARY:
Routinely collected data will be used to assess the morbidity and mortality of cancer patients following a positive COVID-19 infection.

DETAILED DESCRIPTION:
The SARS-CoV-2, (COVID-19) virus of the coronavirus family is believed to have been transmitted from animal to human. On 12th March 2020, the World Health Organisation (WHO) declared this particular coronavirus outbreak a pandemic.

How COVID-19 affects people is still not widely understood. Some people who have tested positive for the virus have been asymptomatic while others, who were otherwise well and healthy before infection, have died. Currently, information obtained so far suggests that most COVID-19 illness, however older people and people with severe comorbidities such as heart and lung disease and diabetes, seem to be at higher risk of developing serious COVID-19 illness.

This research is a retrospective, non-interventional study whose aim is to describe the features of COVID-19 infection specifically in cancer patients; to investigate its severity in this particular population and evaluate the long-term outcomes by means of medical charts review of consecutive patients co-diagnosed with SARS-CoV-2 infection and malignancy.

Patients will be identified from electronic medical records and entered into a pre-designed database. All information used will have been previously collected as part of routine standard of care and will involve but is not limited to: blood test results, prior and current anti-cancer therapy, medical history and most importantly clinical outcomes, such as response to any treatment provided for COVID-19 and patients' survival in relation to baseline clinic-pathologic profile. All data will be collected by each patient's team and will be anonymised and stored in a password-protected NHS computer.

ELIGIBILITY:
Inclusion Criteria:

The investigators will evaluate and include consecutive patients observed in the outpatients and inpatients facility of the study centre meeting all the following CRITERIA:

1. Be ≥18 years of age.
2. Have a confirmed diagnosis of malignancy of any type.
3. Have a confirmed diagnosis of SARS-CoV-2 infection.

Exclusion Criteria:

Patients will not be entered in the study database when one or more of the following CRITERIA are present:

1. Unconfirmed diagnosis of SARS-CoV-2 infection
2. Insufficient clinical/follow up data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients 18 years old or above with cancer and who have also tested positive for Sars-Cov2.
Sampling Method: Non-Probability Sample
Enrollment: 3820 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Describe presenting characteristics and severity or SARS-CoV-2 infection in patients with cancer | 2 years
  Compiling a list of symptoms experienced by patients recruited onto the trial
Assessing what factors are involved in prognosis of cancer patients with COVID-19 | 2 years
  Evaluate prognostic factors for survival in patients with SARS-CoV-2 infection and cancer

CONTACTS AND LOCATIONS:
Overall Officials: David J Pinato, MD, Principal Investigator — Clinical Senior Lecturer and Consultant in Medical Oncology
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cortellini A, Tabernero J, Mukherjee U, Salazar R, Sureda A, Maluquer C, Ferrante D, Bower M, Sharkey R, Mirallas O, Plaja A, Cucurull M, Mesia R, Dalla Pria A, Newsom-Davis T, Van Hemelrijck M, Sita-Lumsden A, Apthorp E, Vincenzi B, Di Fazio GR, Tonini G, Pantano F, Bertuzzi A, Rossi S, Brunet J, Lambertini M, Pedrazzoli P, Biello F, D'Avanzo F, Lee AJX, Shawe-Taylor M, Rogers L, Murphy C, Cooper L, Andaleeb R, Khalique S, Bawany S, Ahmed S, Carmona-Garcia MC, Fort-Culillas R, Linan R, Zoratto F, Rizzo G, Perachino M, Doonga K, Gaidano G, Bruna R, Patriarca A, Martinez-Vila C, Perez Criado I, Giusti R, Mazzoni F, Antonuzzo L, Santoro A, Parisi A, Queirolo P, Aujayeb A, Rimassa L, Diamantis N, Bertulli R, Fulgenzi CAM, D'Alessio A, Ruiz-Camps I, Saoudi-Gonzalez N, Garcia Illescas D, Medina I, Fox L, Gennari A, Aguilar-Company J, Pinato DJ; OnCovid study group. SARS-CoV-2 omicron (B.1.1.529)-related COVID-19 sequelae in vaccinated and unvaccinated patients with cancer: results from the OnCovid registry. Lancet Oncol. 2023 Apr;24(4):335-346. doi: 10.1016/S1470-2045(23)00056-6. Epub 2023 Mar 7. PMID 36898391
- [Derived] Tagliamento M, Gennari A, Lambertini M, Salazar R, Harbeck N, Del Mastro L, Aguilar-Company J, Bower M, Sharkey R, Dalla Pria A, Plaja A, Jackson A, Handford J, Sita-Lumsden A, Martinez-Vila C, Matas M, Miguel Rodriguez A, Vincenzi B, Tonini G, Bertuzzi A, Brunet J, Pedrazzoli P, D'Avanzo F, Biello F, Sinclair A, Lee AJX, Rossi S, Rizzo G, Mirallas O, Pimentel I, Iglesias M, Sanchez de Torre A, Guida A, Berardi R, Zambelli A, Tondini C, Filetti M, Mazzoni F, Mukherjee U, Diamantis N, Parisi A, Aujayeb A, Prat A, Libertini M, Grisanti S, Rossi M, Zoratto F, Generali D, Saura C, Lyman GH, Kuderer NM, Pinato DJ, Cortellini A. Pandemic Phase-Adjusted Analysis of COVID-19 Outcomes Reveals Reduced Intrinsic Vulnerability and Substantial Vaccine Protection From Severe Acute Respiratory Syndrome Coronavirus 2 in Patients With Breast Cancer. J Clin Oncol. 2023 May 20;41(15):2800-2814. doi: 10.1200/JCO.22.01667. Epub 2023 Jan 31. PMID 36720089
- [Derived] Cortellini A, Dettorre GM, Dafni U, Aguilar-Company J, Castelo-Branco L, Lambertini M, Gennatas S, Angelis V, Sita-Lumsden A, Rogado J, Pedrazzoli P, Vinal D, Prat A, Rossi M, Berardi R, Alonso-Gordoa T, Grisanti S, Dimopoulou G, Queirolo P, Pradervand S, Bertuzzi A, Bower M, Arnold D, Salazar R, Tucci M, Harrington KJ, Mazzoni F, Mukherjee U, Tsourti Z, Michielin O, Pommeret F, Brunet J, Vincenzi B, Tonini G, Patriarca A, Biello F, Krengli M, Tabernero J, Pentheroudakis G, Gennari A, Peters S, Romano E, Pinato DJ. Immune checkpoint inhibitor therapy and outcomes from SARS-CoV-2 infection in patients with cancer: a joint analysis of OnCovid and ESMO-CoCARE registries. J Immunother Cancer. 2022 Nov;10(11):e005732. doi: 10.1136/jitc-2022-005732. PMID 36450384
- [Derived] Pinato DJ, Ferrante D, Aguilar-Company J, Bower M, Salazar R, Mirallas O, Sureda A, Bertuzzi A, Brunet J, Lambertini M, Maluquer C, Pedrazzoli P, Biello F, Lee AJX, Sng CCT, Linan R, Rossi S, Carmona-Garcia MC, Sharkey R, Eremiev S, Rizzo G, Bain HD, Yu T, Cruz CA, Perachino M, Saoudi-Gonzalez N, Fort-Culillas R, Doonga K, Fox L, Roldan E, Zoratto F, Gaidano G, Ruiz-Camps I, Bruna R, Patriarca A, Shawe-Taylor M, Fusco V, Martinez-Vila C, Berardi R, Filetti M, Mazzoni F, Santoro A, Delfanti S, Parisi A, Queirolo P, Aujayeb A, Rimassa L, Prat A, Tabernero J, Gennari A, Cortellini A; OnCovid study group. Vaccination against SARS-CoV-2 protects from morbidity, mortality and sequelae from COVID19 in patients with cancer. Eur J Cancer. 2022 Aug;171:64-74. doi: 10.1016/j.ejca.2022.04.036. Epub 2022 May 23. PMID 35704976
- [Derived] Pinato DJ, Aguilar-Company J, Ferrante D, Hanbury G, Bower M, Salazar R, Mirallas O, Sureda A, Plaja A, Cucurull M, Mesia R, Townsend S, Jackson A, Dalla Pria A, Newsom-Davis T, Handford J, Sita-Lumsden A, Apthorp E, Vincenzi B, Bertuzzi A, Brunet J, Lambertini M, Maluquer C, Pedrazzoli P, Biello F, Sinclair A, Bawany S, Khalique S, Rossi S, Rogers L, Murphy C, Belessiotis K, Carmona-Garcia MC, Sharkey R, Garcia-Illescas D, Rizzo G, Perachino M, Saoudi-Gonzalez N, Doonga K, Fox L, Roldan E, Gaidano G, Ruiz-Camps I, Bruna R, Patriarca A, Martinez-Vila C, Cantini L, Zambelli A, Giusti R, Mazzoni F, Caliman E, Santoro A, Grosso F, Parisi A, Queirolo P, Aujayeb A, Rimassa L, Prat A, Tucci M, Libertini M, Grisanti S, Mukherjee U, Diamantis N, Fusco V, Generali D, Provenzano S, Gennari A, Tabernero J, Cortellini A; OnCovid study group. Outcomes of the SARS-CoV-2 omicron (B.1.1.529) variant outbreak among vaccinated and unvaccinated patients with cancer in Europe: results from the retrospective, multicentre, OnCovid registry study. Lancet Oncol. 2022 Jul;23(7):865-875. doi: 10.1016/S1470-2045(22)00273-X. Epub 2022 Jun 2. PMID 35660139
- [Derived] Pinato DJ, Tabernero J, Bower M, Scotti L, Patel M, Colomba E, Dolly S, Loizidou A, Chester J, Mukherjee U, Zambelli A, Dalla Pria A, Aguilar-Company J, Ottaviani D, Chowdhury A, Merry E, Salazar R, Bertuzzi A, Brunet J, Lambertini M, Tagliamento M, Pous A, Sita-Lumsden A, Srikandarajah K, Colomba J, Pommeret F, Segui E, Generali D, Grisanti S, Pedrazzoli P, Rizzo G, Libertini M, Moss C, Evans JS, Russell B, Harbeck N, Vincenzi B, Biello F, Bertulli R, Linan R, Rossi S, Carmona-Garcia MC, Tondini C, Fox L, Baggi A, Fotia V, Parisi A, Porzio G, Saponara M, Cruz CA, Garcia-Illescas D, Felip E, Roque Lloveras A, Sharkey R, Roldan E, Reyes R, Earnshaw I, Ferrante D, Marco-Hernandez J, Ruiz-Camps I, Gaidano G, Patriarca A, Bruna R, Sureda A, Martinez-Vila C, Sanchez de Torre A, Cantini L, Filetti M, Rimassa L, Chiudinelli L, Franchi M, Krengli M, Santoro A, Prat A, Van Hemelrijck M, Diamantis N, Newsom-Davis T, Gennari A, Cortellini A; OnCovid study group. Prevalence and impact of COVID-19 sequelae on treatment and survival of patients with cancer who recovered from SARS-CoV-2 infection: evidence from the OnCovid retrospective, multicentre registry study. Lancet Oncol. 2021 Dec;22(12):1669-1680. doi: 10.1016/S1470-2045(21)00573-8. Epub 2021 Nov 3. PMID 34741822

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT04393974/Prot_SAP_000.pdf